CLINICAL TRIAL: NCT04245371
Title: A Prospective, Randomized, Double-Blind, Cross-over Study of Lidocaine Patch 1.8% in Patients With Moderate to Severe Pain From Carpal Tunnel Syndrome
Brief Title: Lidocaine Patch 1.8% for Moderate to Severe Pain From Carpal Tunnel Syndrome
Acronym: CTS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: John Papakonstantinou, MD (Other)
Collaborators: Scilex Ltd. (Industry)
Responsible Party: Sponsor-Investigator, John Papakonstantinou, MD, Orthopaedic Surgeon, Hand and Upper Extremity Surgeon, Michigan Orthopaedic & Spine Surgeons
Organization: Michigan Orthopaedic & Spine Surgeons (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CTS2020
Record Dates: First submitted 2020-01-22; First posted 2020-01-28 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will serve as their own control
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Active Comparator): Lidocaine Patch 1.8% applied to affected hand at night for 2 weeks following FDA approved dosing recommendations, i.e. 12 hours during each 24-hour daily cycle.
  Interventions: Drug: Lidocaine 1.8%
- Placebo (Placebo Comparator): Placebo Patch applied to affected hand at night for 2 weeks for 12 hours during each 24-hour daily cycle.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine 1.8% — Topical Patch
  Arms: Active
Drug: Placebo — Matching Placebo Patch
  Arms: Placebo

SUMMARY:
The primary objective is to determine the efficacy of Lidocaine Patch 1.8% in reducing the severity of symptoms in participants with moderate-to-severe pain from Carpal Tunnel Syndrome.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, cross-over study. Following informed consent, participants fulfilling entry criteria will be randomly assigned into one of two treatment cohorts. Cohort 1 will be treated with active lidocaine study patch for 1 week following FDA approved dosing recommendations, i.e. 12 hours during each 24-hour daily cycle. Following a 1-week washout period, provided participants continue to meet criteria to proceed, they will then be treated with a placebo topical patch for 1 week. A final visit after another 1-week washout period will complete the study. Participants assigned to the Cohort 2 will be evaluated in the same way except they will enter the placebo arm first and then, after 1-week washout, they will enter the active treatment arm, provided to continue to meet criteria to proceed.

For all measures, participants will serve as their own matched control. Comparisons will be made between significant improvements on active versus placebo treatment arms. The first two-week treatment period is Arm 1; the second two-week period is considered the cross-over arm.

Participants failing treatment will be offered standard of care treatment of steroid injection. All participants will wear a brace for the duration of the study per standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria to be eligible for enrollment into the study:

* Male and female participants, 18 years or older at Screening;
* Participants with Carpal Tunnel Syndrome, confirmed by CT6;
* Pain score of at least 4, based on an 11-point numeric rating scale (NRS) (scale of 0-10), at the screening (baseline) visit;
* Able and willing to provide a written informed consent;
* Able and willing to follow study instructions;
* Able and willing to return to clinic for follow-up visits;
* Able and willing to complete a daily diary;
* Intact skin over the affected wrist;
* Woman of childbearing age agreeing to use 2 forms of contraception.

Exclusion Criteria:

Participants presenting with any of the following exclusion criteria will not be enrolled into the study

* Participants must NOT have had prior steroid injection for CTS, CTS surgery, or other intervention/injury to the wrist that might interfere with assessments in the previous 30 days;
* Participants must not have pain at other sites that interfere with their ability to report site-specific pain related to the study (bilateral CT is an exclusion);
* Participants must NOT have cognitive or psychological impairment that interferes with the ability to complete study related assessments;
* Participants with mild (NRS less than 4) or no pain (only numbness) at baseline prior to randomization;
* Opioid tolerance (receiving at least 1 week of oral morphine 60 mg/day OR transdermal fentanyl 25 mcg/hour OR oral oxycodone 30 mg/day OR oral hydromorphone 8 mg/day OR an equianalgesic dose of any other opioid);
* History of sensitivity or allergy to lidocaine or ZTLIDO;
* Irritated, abraded, or otherwise non-intact skin over the affected wrist;
* Concurrently taking tocainide, mexiletine, or local anesthetics;
* Participants with history of or at significant risk for methemoglobinemia;
* Participation in another study of investigational drugs or devices within 30 days before screening, or previous participation in a Lidocaine Patch study;
* Known to or suspected of not being able to comply with the study protocol;
* Any clinically significant condition that would, in the investigator's opinion, preclude study participation for instance alcohol, medication or drug dependency, neurotic personality, psychiatric illness, epilepsy or suicide risk;
* Pregnancy or nursing mother;
* Woman in childbearing age without satisfactory contraception;
* Presence of possible other cause/s for hand pain (i.e., radicular pain, arthritis, injury, surgery) that could confound assessment or self-evaluation of the pain due to Carpal Tunnel Syndrome;
* Participants using topically applied analgesic compounds on the affected area;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2023-05-07 (Actual); Study Completion 2023-05-07 (Actual)

PRIMARY OUTCOMES:
Symptom Severity Scale (SSS) of the Boston Carpal Tunnel Questionnaire (BCTQ): minimally clinically important difference | After 1 Week of Treatment
  The minimum score is 11 indicating low symptom severity and the maximum score is 55 which would indicate high symptom severity.

SECONDARY OUTCOMES:
Functional Status Score (FSS) of the Boston Carpal Tunnel Questionnaire (BCTQ):minimally clinically important difference | After 1 Week of Treatment
  The minimum score is 8 indicating low symptom severity and the maximum score is 40 which would indicate high symptom severity.
Sensory examination | After 1 Week of Treatment
  Clinical sensory neurological examination will assess for response to light touch, pinprick, and vibration.
Pain Detect Questionnaire | After 1 Week of Treatment
  The Pain DETECT questionnaire screens for components of neuropathic pain: intensity, pattern and quality.

CONTACTS AND LOCATIONS:
Overall Officials: John Papakonstantinou, MD, Principal Investigator — Michigan Orthopaedic & Spine Surgeons
Locations (1):
- Michigan Orthopaedic & Spine Surgeons, Rochester Hills, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chung SY, Kwak JM, Kang S, Son SH, Kim JD, Yoon JS. Predictive Variables for Sonographically Guided Corticosteroid Injection in Mild-to-Moderate Carpal Tunnel Syndrome. Ann Rehabil Med. 2018 Apr;42(2):213-221. doi: 10.5535/arm.2018.42.2.213. Epub 2018 Apr 30. PMID 29765874
- [Background] Chesterton LS, Blagojevic-Bucknall M, Burton C, Dziedzic KS, Davenport G, Jowett SM, Myers HL, Oppong R, Rathod-Mistry T, van der Windt DA, Hay EM, Roddy E. The clinical and cost-effectiveness of corticosteroid injection versus night splints for carpal tunnel syndrome (INSTINCTS trial): an open-label, parallel group, randomised controlled trial. Lancet. 2018 Oct 20;392(10156):1423-1433. doi: 10.1016/S0140-6736(18)31572-1. PMID 30343858
- [Background] Moghtaderi AR, Jazayeri SM, Azizi S. EMLA cream for carpal tunnel syndrome: how it compares with steroid injection. Electromyogr Clin Neurophysiol. 2009 Sep-Oct;49(6-7):287-9. PMID 19845100
- [Background] Leppert W, Malec-Milewska M, Zajaczkowska R, Wordliczek J. Transdermal and Topical Drug Administration in the Treatment of Pain. Molecules. 2018 Mar 17;23(3):681. doi: 10.3390/molecules23030681. PMID 29562618
- [Background] Sears ED, Meerwijk EL, Schmidt EM, Kerr EA, Chung KC, Kamal RN, Harris AHS. Variation in Nonsurgical Services for Carpal Tunnel Syndrome Across a Large Integrated Health Care System. J Hand Surg Am. 2019 Feb;44(2):85-92.e1. doi: 10.1016/j.jhsa.2018.11.002. Epub 2018 Dec 20. PMID 30579690
- [Background] Okamura A, Guidetti BC, Caselli R, Borracini JA, Moraes VY, Belloti JC. HOW DO BOARD-CERTIFIED HAND SURGEONS MANAGE CARPAL TUNNEL SYNDROME? A NATIONAL SURVEY. Acta Ortop Bras. 2018 Jan-Feb;26(1):48-53. doi: 10.1590/1413-785220182601181880. PMID 29977145
- [Background] Graham B. The value added by electrodiagnostic testing in the diagnosis of carpal tunnel syndrome. J Bone Joint Surg Am. 2008 Dec;90(12):2587-93. doi: 10.2106/JBJS.G.01362. PMID 19047703
- [Background] Aroori S, Spence RA. Carpal tunnel syndrome. Ulster Med J. 2008 Jan;77(1):6-17. PMID 18269111
- See also: FULL PRESCRIBING INFORMATION of ZTLIDO (lidocaine topical system) 1.8% — https://www.accessdata.fda.gov/drugsatfda_docs/label/2018/207962s000lbl.pdf